CLINICAL TRIAL: NCT06726746
Title: Efficacy of Fractional CO2 Laser Treatment in Post-Menopausal Women With Vaginal Atrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Daniel Onsi Anis, Dr, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Post Menopausal Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention by using the Fractional CO2 laser (Experimental): . Using the following settings with the internal handpiece: square pattern with Deep Mode, fractional density of 5% and energy level of 50 mJ and fluence of 283 J/cm2. The handpiece will be inserted into the vagina (up to 10 cm) The handpiece will be positioned with contact to the vagina and will be rotated to apply 12 pulses at each 1-cm marking (application of laser energy at 3-10-cm depths) until the distal end of the vaginal probe reaches the introitus.
  The laser application will be performed on an outpatient basis without local anesthesia in outpatient clinic.
  Interventions: Device: Fractional CO2 laser

INTERVENTIONS:
Device: Fractional CO2 laser — . Using the following settings with the internal handpiece: square pattern with Deep Mode, fractional density of 5% and energy level of 50 mJ and fluence of 283 J/cm2. The handpiece will be inserted into the vagina (up to 10 cm) The handpiece will be positioned with contact to the vagina and will be rotated to apply 12 pulses at each 1-cm marking (application of laser energy at 3-10-cm depths) until the distal end of the vaginal probe reaches the introitus.
  The laser application will be performed on an outpatient basis without local anesthesia in outpatient clinic.

SUMMARY:
Vaginal dryness, itching, burning, irritability, secretion, and various urinary problems are the symptoms of vulvovaginal atrophy. Therefore, more attention must be paid to relieve these symptoms in order to provide better sexual health for postmenopausal women. At present, an accumulating body of evidence suggests safety and efficacy of laser and energy-based devices for the treatment of women's genitourinary conditions. More clinical studies are needed to assess the safety profile and clinical outcomes of the lasers and energy-based devices to treat the symptoms associated with vulvovaginal atrophy (VVA)

DETAILED DESCRIPTION:
This is a prospective, investigational study that will be performed in private outpatient clinic on 30 participants.

All participants will be scheduled for four visits (V1, V2, V3, and V4) with a 4- week interval where they will receive the interventions in the first three visits (V1, V2, and V3), While in the last visit (V4), the study will assess the participants' satisfaction with the treatment and any adverse events they experienced during the study period.

Detailed medical history of all participants will be collected including age, age at menopause, parity, type of delivery, history of vaginal reconstructive surgery, history of hormonal treatment, and sexual activity status.

At each visit (V1, V2, V3, and V4), the participants will be interviewed to assess Vaginal Health Index using the VHI score and assess the changes in the Female Sexual Function Index FSFI.

Signs of vaginal atrophy will be evaluated during pelvic examination After pelvic examination and completion of the questionnaire, the interventions will be performed.

The participants will receive the interventions in the first three visits (V1, V2, and V3).While in the last visit (V4), the study will assess the participants' satisfaction with the treatment and any adverse events they experienced during the study period.

The Procedures will be performed in private outpatient clinic. The participants will receive the intervention by using the CO2 laser machine. Using the following settings with the internal handpiece: square pattern with Deep Mode, fractional density of 5% and energy level of 50 mJ and fluence of 283 J/cm2. The handpiece will be inserted into the vagina (up to 10 cm) The handpiece will be positioned with contact to the vagina and will be rotated to apply 12 pulses at each 1-cm marking (application of laser energy at 3-10-cm depths) until the distal end of the vaginal probe reaches the introitus.

The laser application will be performed on an outpatient basis without local anesthesia in outpatient clinic.

Participants will be advised to avoid sexual intercourse or intravaginal devices for at least 3 days after the procedure owing to transient local inflammation at the vaginal mucosa generated by the laser application.

ELIGIBILITY:
Inclusion Criteria:

1. Menopausal women whose ages ranged from 45 to 65 years.
2. Sexually active
3. Had symptoms of VVA (vaginal dryness, irritation, soreness, or dyspareunia)

Exclusion Criteria:

1. Any history of hormonal therapy within the past 6 months
2. Vaginal moisturizer or lubricant applications within the past 30 days
3. Acute/recurrent urinary tract infection
4. Active genital infection
5. Prolapse stage II or more based on examination
6. Psychiatric disorders
7. Undiagnosed vaginal bleeding
8. Any serious disease or chronic condition that could interfere with study compliance

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The Vulvovaginal Symptoms Questionnaire (VVSQ) | 4-6 months
The Vaginal Health Index VHI assessment. | 4-6 months

SECONDARY OUTCOMES:
Urogenital Distress Short Form (UDI-6 | 4-6 months
Incontinence Impact Questionnaire Short Form (IIQ-7) | 4-6 months
Female Sexual Function Index (FSFI) | 4-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided